CLINICAL TRIAL: NCT00726193
Title: A Prospective Randomized Multi - Center Clinical Outcomes Collection Study To Analyze The Effect Of Ebi Osteogen™ Direct Current Stimulator On The Surgical Reconstruction Of Tibia Nonunions
Brief Title: Study to Analyze the Effects of EBI OsteoGen™ on the Surgical Reconstruction of Tibia Non-unions
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment, lack of follow up
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-012
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Tibia Fracture Non Union Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 - standard films: Tibia reconstruction surgery with OsteoGen™ with standard radiographs
  Interventions: Device: OsteoGen
- 2 - Standard films plus CT: Tibia reconstruction surgery with OsteoGen™ with standard radiographs and additional CT scan at 10 and 18 weeks.
  Interventions: Device: OsteoGen

INTERVENTIONS:
Device: OsteoGen — OsteoGen Implatable stimulator

SUMMARY:
The purpose of this clinical outcomes collection study is to analyze the effect of the EBI OsteoGen™ Direct Current Stimulator upon surgical reconstruction of tibia nonunion (no visible progressive signs of healing) fracture in a prospective database.

DETAILED DESCRIPTION:
This clinical outcomes collection study is to analyze the effect of the EBI OsteoGen™ Direct Current Stimulator upon surgical reconstruction of tibia nonunion (no visible progressive signs of healing) fracture in a prospective database.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of a tibia nonunion.
2. Male or female between ages of 18 and 75 years old, inclusive

Exclusion Criteria:

1. Subject has open wounds or underlying osteomyelitis.
2. Subject has associated multiple traumas, and/or fractures that are not anatomically reduced or lose reduction at later time points.
3. If female, subject is pregnant, plans on becoming pregnant during the duration of this clinical outcomes collection study or lactating.
4. Subject has an implanted unipolar pacemaker.
5. Subject has active cancer.
6. Subject has severe peripheral vascular disease (ABI <0.4)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: private practice patients
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2006-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for this trial will be the percentage of successful tibia unions achieved | 8 Months

SECONDARY OUTCOMES:
Mean AOFAS Score (% Change From Baseline), Foot Function Index (% Change from Baseline), SF-36 Health Survey (Change from Baseline) | 8 Months

CONTACTS AND LOCATIONS:
Overall Officials: Joel Batts, Study Director — Biomet Spine
Locations (1):
- Orthopedic Foot and Ankle Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided